CLINICAL TRIAL: NCT01893619
Title: Observational Research on Use of Immunoprop Supplement in Chronic Fatigue Syndrome
Acronym: immunoprop
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York CFS Association (Other)
Responsible Party: Sponsor
Other Study IDs: immunoprop
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue syndrome; Karnofsky score; supplements
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Observational study regarding the use of supplements in chronic fatigue syndrome patients

DETAILED DESCRIPTION:
Detailed questionnaire regarding the diagnosis of an onset of chronic fatigue syndrome and 100 patients. using Karnofsky scale before and after use of supplements patient scores are compared in a double blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Fukuda criteria and Canadian consensus criteria will be the diagnosis criteria for patient selection

Exclusion Criteria:

* non inclusion in the above criteria

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fukuda criteria and Canadian consensus criteria will be the diagnosis criteria for patient selection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Karnovsky score comparison | Six months
  Review of Karnofsky score over prior to diagnosis and subsequent to patients having taken supplements

CONTACTS AND LOCATIONS:
Overall Officials: DEREK enlander, Principal Investigator — CFIDS RESEARCH FOUNDATION
Locations (1):
- Me/Cfs Center,860 Fifth Avenue, New York, New York, United States